CLINICAL TRIAL: NCT03340961
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group, Controlled Study to Assess the Efficacy, Safety and Tolerability of Oral DFD-29 Extended Release Capsules for the Treatment of Inflammatory Lesions of Rosacea Over 16 Weeks
Brief Title: A Controlled Study to Assess the Efficacy, Safety and Tolerability of Oral DFD-29 Extended Release Capsules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFD-29-CD-002
Record Dates: First submitted 2017-10-19; First posted 2017-11-14 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Doxycycline; Capsules

STUDY DESIGN:
Intervention Model Description: A Multi-Center, Randomized, Double-Blind, Parallel-Group, Controlled Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each subject will be allocated to one of the following treatment groups, receiving 1 capsule once daily in the morning for 16 weeks:
  1. DFD-29 Extended Release Capsules (40 mg)
  2. DFD-29 Extended Release Capsules (20 mg)
  3. Doxycycline Modified Release Hard Capsules (40 mg)
  4. Placebo Capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DFD-29 Extended Release Capsules (40 mg) (Experimental): DFD-29 (minocycline HCl) Extended Release Capsules (40 mg) once per day for 16 weeks.
  Interventions: Drug: DFD-29 Extended Release Capsules (40 mg)
- DFD-29 Extended Release Capsules (20 mg) (Experimental): DFD-29 (minocycline HCl) Extended Release Capsules (20 mg) once per day for 16 weeks.
  Interventions: Drug: DFD-29 Extended Release Capsules (20 mg)
- Oraycea® (doxycycline) Capsules (Experimental): Oraycea® (doxycycline) Modified Release Hard Capsules (40 mg) once per day for 16 weeks.
  Interventions: Drug: Oraycea® (doxycycline) Capsules
- Placebo Capsules (Placebo Comparator): Placebo Capsules once per day for 16 weeks.
  Interventions: Drug: Placebo Capsules

INTERVENTIONS:
Drug: DFD-29 Extended Release Capsules (40 mg) — Oral Treatment
  Arms: DFD-29 Extended Release Capsules (40 mg)
Drug: DFD-29 Extended Release Capsules (20 mg) — Oral Treatment
  Arms: DFD-29 Extended Release Capsules (20 mg)
Drug: Oraycea® (doxycycline) Capsules — Oral Treatment
  Arms: Oraycea® (doxycycline) Capsules
Drug: Placebo Capsules — Oral Treatment
  Arms: Placebo Capsules

SUMMARY:
Clinical assessments of efficacy will be conducted based on Investigator's Global Assessment (IGA, modified scale without erythema), Clinician's Erythema Assessment (CEA), and on inflammatory lesion counts at Weeks 4, 8, 12 and 16 in comparison to Baseline.

DETAILED DESCRIPTION:
Two hundred (200) male and female subjects with papulopustular rosacea will be enrolled to get 176 completed subjects (forty-four (44) completers each in groups 1 to 4).

After assessing eligibility during an up to 28 days screening period, 200 subjects will be enrolled in the study (fifty subjects each in groups 1 to 4). Subject visits are scheduled at Screening, Baseline (Day 1), and Weeks 4, 8, 12 and 16.

Clinical assessments of efficacy will be conducted based on Investigator's Global Assessment (IGA, modified scale without erythema), Clinician's Erythema Assessment (CEA), and on inflammatory lesion counts at Weeks 4, 8, 12 and 16 in comparison to Baseline. Additionally, high sensitivity C-reactive protein (hs-CRP) in the blood will be assessed at Baseline, and at Week 16 to explore any impact of the treatment on the inflammatory pathology.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to understand the requirements of the study and be willing to give written informed consent.
2. Male and female subjects aged 18 years and above.
3. Subjects, any gender or ethnicity (and of Fitzpatrick skin type I - III), must be in good general health as determined by the Investigator.
4. Subjects must have a clinical diagnosis of papulopustular rosacea, IGA grade 2 - 4.
5. Subjects must have 10 - 40 (both inclusive) inflammatory lesions (papules and pustules) of rosacea over the face.
6. Subjects must have not more than 2 nodules.
7. Subjects with moderate to severe erythema with a total score of 5 - 20 on the CEA scale.
8. Females must have a negative urine pregnancy test at the screening and baseline visit.
9. Females must either be postmenopausal with no menses for at least 12 months or surgically sterile (hysterectomy or tubal ligation) or agree to use a highly effective method of contraception with a pearl index of <1% up to 1 month after last dose.
10. Subjects must be in good general health as determined by the investigator and supported by the medical history and normal or not clinically significant abnormal vital signs (blood pressure and pulse).

Exclusion Criteria:

1. Females who are pregnant or nursing or planning to become pregnant during the study.
2. Male whose female partner is planning to conceive a child.
3. Subjects who have been treated for rosacea within the 30 days prior to the Baseline Visit (e.g. metronidazole, azelaic acid, doxycycline or brimonidine).
4. Subjects who have been treated with systemic retinoids within 6 months prior to the Baseline visit.
5. Subjects who have participated in a trial involving any investigational product in the 90 days prior to the Baseline Visit.
6. Subjects with any disease or medical condition that would interfere with the study outcome or place the subject at undue risk.
7. Subjects who use or have used systemic steroids within the 30 days prior to the Baseline Visit or any other immunosuppressive medication.
8. Subjects who are on anti-coagulants or those who are likely to require anti-coagulants during the study period.
9. History of drug or alcohol abuse in the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sidgiddi, MD, Study Director — Director-Clinical Development
Locations (14):
- Germany (14):
  - Site 13, Bad Bentheim
  - Site 07, Berlin
  - Site 14, Berlin
  - Site 09, Bochum
  - Site 05, Buxtehude
  - Site 15, Darmstadt
  - Site 03, Dülmen
  - Site 08, Leipzig
  - Site 11, Mahlow
  - Site 06, Münster
  - Site 10, Osnabrück
  - Site 01, Pommelsbrunn
  - Site 04, Potsdam
  - Site 02, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsianakas A, Pieber T, Baldwin H, Feichtner F, Alikunju S, Gautam A, Shenoy S, Singh P, Sidgiddi S. Minocycline Extended-Release Comparison with Doxycycline for the Treatment of Rosacea: A Randomized, Head-to-Head, Clinical Trial. J Clin Aesthet Dermatol. 2021 Dec;14(12):16-23. PMID 35096250

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DFD-29 Extended Release Capsules (40 mg) | DFD-29 Extended Release Capsules (20 mg) | Oraycea® (Doxycycline) Capsules | Placebo Capsules
Started | 53 | 50 | 49 | 53
Completed | 47 | 38 | 40 | 35
Not Completed | 6 | 12 | 9 | 18
Not completed — Adverse Event | 1 | 3 | 2 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 4 | 7
Not completed — Use of prohibited treatment | 0 | 3 | 2 | 4
Not completed — Wrongful enrollment (I/E criteria not me | 0 | 1 | 0 | 1
Not completed — Subject developed an exclusion criterion | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The FAS (full analysis set) had all subjects who had at least one post Baseline efficacy assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | DFD-29 Extended Release Capsules (40 mg) | DFD-29 Extended Release Capsules (20 mg) | Oraycea® (Doxycycline) Capsules | Placebo Capsules | Total
Number analyzed (Participants) | 53 | 50 | 49 | 53 | 205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 40 | 40 | 42 | 167
  >=65 years | 8 | 10 | 9 | 11 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (15.05) | 51.1 (13.13) | 51.6 (12.94) | 52.5 (12.92) | 50.5 (13.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 29 | 27 | 124
  Male | 19 | 16 | 20 | 26 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 53 | 50 | 49 | 53 | 205
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 53 | 50 | 49 | 53 | 205
Total Inflammatory Lesion Count [Mean (Standard Deviation); unit: Number of lesions] | 23.8 (8.69) | 24.5 (9.49) | 23.8 (7.56) | 24.0 (8.40) | 24.0 (8.51)

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment (IGA) 0=Clear, 1=Near Clear, 2=Mild, 3=Moderate, 4=Severe
Description: Proportion of subjects with Investigator Global Assessment (IGA) 'treatment success' - Grade 0 or 1 at the end of study with at least 2 grade reduction from Baseline to Week 16.
Time Frame: 16 weeks
Population: The FAS (full analysis set) included all subjects that had at least one post Baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DFD-29 Extended Release Capsules (40 mg) | DFD-29 Extended Release Capsules (20 mg) | Oraycea® (Doxycycline) Capsules | Placebo Capsules
Number analyzed (Participants) | 53 | 47 | 48 | 52
Participants | 35 | 15 | 16 | 6

2. Primary Outcome: Total Inflammatory Lesion Count Reduction
Description: The total inflammatory lesion count is carried out by visual inspection by the Investigator at every study visit from Screening up to Week 16 (or at early termination). Inflammatory lesions will be recorded on a diagram of a human face, divided in 4 quadrants.
Time Frame: 16 Weeks
Population: FAS population
Measure: Mean (Standard Deviation); unit: Count of lesions
Arm/Group | DFD-29 Extended Release Capsules (40 mg) | DFD-29 Extended Release Capsules (20 mg) | Oraycea® (Doxycycline) Capsules | Placebo Capsules
Number analyzed (Participants) | 53 | 47 | 48 | 52
Count of lesions | -19.2 (9.72) | -12.6 (12.92) | -10.5 (15.18) | -7.3 (10.12)

3. Secondary Outcome: Median Change in RosaQoL (Rosacea Quality of Life) Score From Baseline to Week 16
Description: The RosaQoL assessment is carried out by the Investigator using the validated RosaQoL questionnaire, at every study visit from Screening up to Week 16 (or at early termination). The RosaQol tool has 21 questions related to the impact that Rosacea has on various dimensions influencing quality of life. Each question is graded from 1 (Never) - 5 (All the time), thus leading to a minimum score of 21 (21 x 1) to a maximum score of 105 (21 x 5) per subject at every visit. Higher the score, poorer is the quality of life. This outcome measured the change in the score from Baseline to Week 16.
Time Frame: Median change in the score from Baseline to Week 16
Population: FAS Population
Measure: Median (Full Range); unit: score on a scale
Arm/Group | DFD-29 Extended Release Capsules (40 mg) | DFD-29 Extended Release Capsules (20 mg) | Oraycea® (Doxycycline) Capsules | Placebo Capsules
Number analyzed (Participants) | 53 | 47 | 48 | 52
score on a scale | -11.0 [-53 to 11] | -8.0 [-34 to 8] | -3.0 [-30 to 25] | -1.0 [-37 to 19]

ADVERSE EVENTS:
Time Frame: AEs were collected from subjects from the time of signing of the ICF up to Week 16/End of Study Visit.
Description: Adverse events were collected by spontaneous reports from subjects, either verbal or recorded in the subject's diary, by directed question of subjects, and by observation. All AEs from the time of signing of the ICF up to the EOS visit were recorded.
  AEs occurring from the time of first study drug administration up to the End-of-Study were defined as treatment emergent AEs.
Arm/Group | DFD-29 Extended Release Capsules (40 mg) | DFD-29 Extended Release Capsules (20 mg) | Oraycea® (Doxycycline) Capsules | Placebo Capsules
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/48 | 0/48 | 0/53
Serious Adverse Events (participants affected / at risk) | 1/52 | 2/48 | 2/48 | 0/53
Other Adverse Events (participants affected / at risk) | 37/52 | 33/48 | 27/48 | 35/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-29 Extended Release Capsules (40 mg) (N=52) | DFD-29 Extended Release Capsules (20 mg) (N=48) | Oraycea® (Doxycycline) Capsules (N=48) | Placebo Capsules (N=53)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Coronary artery disease
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Atrial fibrillation
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Lymphoma
Papilloma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Papilloma
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Retinal detachment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DFD-29 Extended Release Capsules (40 mg) (N=52) | DFD-29 Extended Release Capsules (20 mg) (N=48) | Oraycea® (Doxycycline) Capsules (N=48) | Placebo Capsules (N=53)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (9) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 4 (4) | 0 (0) | 3 (7)
Nasopharyngitis (Investigations) | 11 (11) | 8 (11) | 7 (7) | 6/35 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 4 (6) | 6 (6)
Headache (Nervous system disorders) | 22 (47) | 14 (35) | 13 (37) | 13 (29)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT03340961/SAP_000.pdf
  • Study Protocol (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT03340961/Prot_001.pdf